CLINICAL TRIAL: NCT04210219
Title: A Phase 1, Open-Label Study of the Safety, Pharmacokinetics, and Pharmacodynamics of JNJ-64264681 in Participants With Non-Hodgkin Lymphoma and Chronic Lymphocytic Leukemia
Brief Title: A Study of JNJ-64264681 in Participants With Non-Hodgkin Lymphoma and Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CR108706; 64264681LYM1001 (Other: Janssen Research & Development, LLC); 2019-003194-25 (EudraCT Number); 2024-512686-13-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2019-12-23; First posted 2019-12-24 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Lymphoma, Non-Hodgkin; Leukemia, Lymphocytic, Chronic, B-Cell
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — JNJ-64264681

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- JNJ-64264681: Dose Escalation and Expansion (Experimental): Participants will receive oral administration of JNJ-64264681 capsule at a dose assigned by the sponsor Study Evaluation Team (SET), based on the available safety, pharmacokinetics, and pharmacodynamics data in dose escalation treatment group (Part 1); and recommended Phase 2 dose (RP2D) determined in Part 1 in cohort expansion treatment group (Part 2).
  Interventions: Drug: JNJ-64264681

INTERVENTIONS:
Drug: JNJ-64264681 — JNJ-64264681 capsule will be administered orally.

SUMMARY:
The purpose of the study is to determine the recommended Phase 2 dose(s) (RP2D[s]) in B cell non-Hodgkin lymphoma (NHL) and chronic lymphocytic leukemia (CLL) in Part 1 and to evaluate the safety of JNJ-64264681 at the RP2D(s) in Part 2.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have Eastern Cooperative Oncology Group (ECOG) performance status grade of 0 or 1
* Participants must have cardiac parameters within the following range: corrected QT interval (QTcF) less than or equal to <= 480 milliseconds based on the average of triplicate assessments performed as close as possible in succession (the full set of triplicates should be completed in less than 10 minutes)
* Women of childbearing potential must have a negative highly sensitive serum pregnancy test (example: beta human chorionic gonadotropin [beta-hCG]) at screening, and a negative serum or urine pregnancy test prior to the first dose of study drug
* Women must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study and for a period of at least 30 days after the last study drug administration
* Participants must be willing and able to adhere to the lifestyle restrictions specified in this protocol

Exclusion Criteria:

* Participant has known active central nervous system (CNS) involvement
* Participant has received prior solid organ transplantation
* Participant has known allergies, hypersensitivity, or intolerance to JNJ-64264681 or its excipients
* Participant has been treated with an investigational drug (including investigational vaccines) within five half-lives or 2 weeks before the planned first dose of study drug
* Participant is experiencing toxicities from previous anticancer therapies that have not resolved to baseline levels, or to Grade 1 or less (except for alopecia and peripheral neuropathy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2020-07-02 (Actual); Primary Completion 2025-05-28 (Actual); Study Completion 2025-05-28 (Actual)

PRIMARY OUTCOMES:
Part 1: Number of Participants With Dose Limiting Toxicity (DLT) | Up to 21 days
  The DLTs are based on drug related adverse events and defined as any of the following events: hematological or non-hematological toxicity of grade 3 or higher (as specified in protocol).
Part 1 and Part 2: Number of Participants with Adverse Events (AEs) | Up to 2 years
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.

SECONDARY OUTCOMES:
Plasma Concentration of JNJ-64264681 | Up to 2 years
  Plasma concentration of JNJ-64264681 will be evaluated.
Percentage Occupancy of the Target | Up to 2 years
  The pharmacodynamics of JNJ-64264681 will be assessed by determining the percentage of target occupancy. Blood samples will be obtained for pharmacodynamic assessments (target occupancy).
Overall Response Rate (ORR) | Up to 2 years
  ORR is defined as the percentage of participants who achieve a complete response (CR) + partial response (PR) or better according to the Revised Response Criteria for Malignant Lymphoma and the International Workshop on Chronic Lymphocytic Leukemia (iwCLL) Response Criteria and International Workshop for Waldenstrom Macroglobulinemia (IWWM) Response Criteria.
Time to Response (TTR) | Up to 2 years
  TTR is defined for participants who achieved PR or CR as the time from the first dose of study drug to first response of PR or CR according to the Revised Response Criteria for Malignant Lymphoma and iwCLL Response Criteria and IWWM Response Criteria.
Duration of Response (DOR) | Up to 2 years
  DOR is defined for participants who achieved PR or CR as the time between the date of initial documentation of PR or CR to the date of either the first documented evidence of disease progression or death according to the Revised Response Criteria for Malignant Lymphoma and iwCLL Response Criteria and IWWM Response Criteria.
Complete Response (CR) Rate | Up to 2 years
  CR rate is defined as the percentage of participants who achieve a best response of CR according to the Revised Response Criteria for Malignant Lymphoma and iwCLL Response Criteria and IWWM Response Criteria.
Progression-free Survival (PFS) | Up to 2 years
  PFS is defined as the time from the date of the first dose of the study drug to the date of either the first documented disease progression (according to the Revised Response Criteria for Malignant Lymphoma and iwCLL Response Criteria and IWWM Response Criteria), or death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (15):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States
- Arensia Exploratory Medicine, Tbilisi, Georgia
- Arensia Exploratory Medicine, Chisinau, Moldova
- Poland (4):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Pratia Onkologia Katowice, Katowice
  - Pratia MCM Krakow, Krakow
  - Centrum Medyczne Pratia Poznan, Skorzewo
- Taiwan (5):
  - Chang-Gung Memorial Hospital, Kaohsiung, Kaohsiung County
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
- Medical Center of Limited Liability Company Arensia Exploratory Medicine, Kyiv, Ukraine
- United Kingdom (2):
  - Queen Mary University of London, Charterhouse Square
  - Plymouth Hospitals NHS Trust, Plymouth

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency